CLINICAL TRIAL: NCT03295786
Title: Phase 1-2, Randomised, Double-Blind, Placebo Controlled, Safety and Tolerability Study of Intraputamenal Cerebral Dopamine Neurotrophic Factor (CDNF) Infusions Via an Investigational Drug Delivery System to Patients With Parkinson's Disease
Brief Title: Clinical Study to Test the Safety of CDNF by Brain Infusion in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Collaborators: Renishaw plc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-CD-CL-2002; 2015-004175-73 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-28 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease; Movement Disorders; Neurodegenerative Diseases; Nervous System Diseases; Brain Diseases
Keywords: Parkinson; CDNF; Drug Delivery System; Intracerebral
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Neurodegenerative Diseases; Nervous System Diseases; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Randomised, Double-Blind, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Patients randomized to this group will receive 6 monthly infusions of placebo/vehicle
  Interventions: Drug: Cerebral Dopamine Neurotrophic Factor; Device: Renishaw Drug Delivery System
- CDNF mid-dose (Experimental): Patients randomized to this group will receive 6 doses of CDNF titrated to mid-dose
  Interventions: Drug: Cerebral Dopamine Neurotrophic Factor; Device: Renishaw Drug Delivery System
- CDNF high-dose (Experimental): Patients randomized to this group will receive 6 doses of CDNF titrated to high-dose
  Interventions: Drug: Cerebral Dopamine Neurotrophic Factor; Device: Renishaw Drug Delivery System

INTERVENTIONS:
Drug: Cerebral Dopamine Neurotrophic Factor — Repeated intracerebral infusions
  Other Names: CDNF
Device: Renishaw Drug Delivery System — Stereotactically implanted device
  Other Names: DDS

SUMMARY:
This study evaluates the safety and tolerability of CDNF in patients with Parkinson's disease, when dosed directly into the brain using an implanted investigational drug delivery system (DDS). Safety and accuracy of the DDS is also being evaluated. One-third of the patients will receive monthly infusions with placebo and two-third of the patients will receive monthly infusions with either mid- or high-doses of CDNF for a period of 6 months.

DETAILED DESCRIPTION:
A patient's participation in the study will last for ten months and will include sixteen to seventeen visits:

* Screening (2 visits)
* Planning of surgery - Surgery: implantation of drug delivery system - Post-surgery follow-up (3 visits)
* Test infusions with vehicle (1-2 visits)
* Positron emission tomography (PET) examinations before the first and after the last dose (2 visits)
* Baseline and randomisation to CDNF or placebo group (1 visit)
* Dosing visits: CDNF or placebo (6 visits)
* End-of-study visit (1 visit)

Study examinations and assessments

- Physical examination: pulse rate, blood pressure, temperature, body weight and height

* ECG (electrocardiography) and blood and urine tests
* HIV, hepatitis B and C blood tests (on first visit)
* Pregnancy tests for women of childbearing age
* Completion of a patient diary to record mobility and time asleep
* Parkinson's Kinetigraph (PKGTM) Data Logger: a watch-type device worn on the wrist for certain periods during the study to record movements
* Questionnaires, rating scales and forms: quality of life, mood, memory, impulse control, mental health
* Assessment of the port and the skin around the port
* Cerebrospinal fluid sampling by lumbar puncture
* Magnetic resonance imaging (MRI)
* Positron emission tomography scans (PET)
* Computed tomography (CT)

For more information: https://treater.eu/clinical-study/

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease based on UK brain bank criteria
2. Duration of PD motor symptoms 5-15 years (inclusive)
3. Age 35-75 years (inclusive)
4. Presence of motor fluctuations.
5. At least 5 daily doses of levodopa
6. Ability to reliably distinguish motor states and accurately complete fluctuation diaries
7. UPDRS motor score (part III) in a practically defined OFF-state between 25-50 (inclusive)
8. Hoehn and Yahr ≤ stage III in the OFF-state
9. Responsiveness to levodopa
10. No change in anti-parkinsonian medication for 6 weeks before screening
11. Provision of Informed Consent

Exclusion Criteria:

1. Diagnosed with atypical parkinsonism or any known secondary parkinsonian syndrome.
2. Signs or symptoms suggestive of atypical parkinsonian syndrome.
3. Drug-resistant rest tremor.
4. Prior neurosurgical treatment for PD, including lesioning or deep brain stimulation
5. Significant neurological disorder other than PD including clinically significant head trauma, cerebrovascular disease, epilepsia, CSF shunt or other implanted CNS device
6. Presence of significant depression as defined as a BDI score ≥ 20
7. Current psychosis requiring therapy.
8. Presence of clinically significant impulse control disorder ((QUIP-RS) score > 20), or, presence of dopamine dysregulation syndrome.
9. MoCA score < 24.
10. Use within 3 months of planned catheter insertion of concomitant medications known to affect PD symptoms other than prescribed PD therapy.
11. Any medical condition, which might impair outcome measure assessments or safety measures including ability to undergo MRI or DAT-PET.
12. Hypersensitivity or allergy to gadolinium or to any of excipients of macrocyclic GBCA used for the surgical planning MRI.
13. Screening and/or planning MRI demonstrating any abnormality, which would suggest an alternative cause for patient's parkinsonism or preclude neurosurgery.
14. Any medical condition that would put the patient at undue risk from surgical treatment or chronic implants including but not limited to bleeding disorders, chronic infections, or immunosuppressive illness
15. History within the last 5 years of cancer with the exception of basal cell carcinoma of the skin
16. History of drug or alcohol abuse within 2 years of screening
17. Use of any investigational drug or device within 90 days of screening
18. Active breastfeeding

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Week 15 to Week 40
  Number and severity of adverse events
Electrocardiogram (ECG) | Week 15 to Week 40
  Changes in electrical activity of heartbeat measured by electrocardiogram
Beck Depression Inventory (BDI) score | Week 15 to Week 40
  Assessment of change in depression using Beck Depression Inventory (BDI) score
Questionnaire for impulsive-compulsive disorder in Parkinson's disease rating scale (QUIP_RS) | Week 15 to Week 40
  Assessment of changes in impulsive-compulsive disorders using QUIP_RS
Montreal cognitive assessment (MoCA) | Week 15 to Week 40
  Assessment of change in cognitive domains using MoCA test
Physical examination | Week 15 to Week 40
  Changes in anatomic findings found in physical examination
Vital signs | Week 15 to Week 40
  Changes in vital signs
Clinical laboratory safety screen | Week 15 to Week 40
  Changes in clinical laboratory variables (chemistry, haematology, urinanalysis)
Formation of anti-CDNF antibodies | Week 15 to Week 40
  Change in anti-CDNF antibody concentration
Device related changes in safety measures | Week 8 to Week 40
  Occurrence of adverse device effects (ADE), for either the whole system or the individual sub systems (guide tubes/catheters, subcutaneous components, port), serious adverse device effect (SADE) including long term effects, neurological deficit (seizures), infection (local to components, in CNS), severe skin breakdown or necrosis requiring component removal life threatening or major (requiring intervention) intracerebral haemorrhage.
Device related accuracy of implantation | Week 8
  The accuracy of implantation of the Drug Delivery System (DDS) will be measured comparing the tip of each individual catheters defined in the plan of the surgical procedure with the position of those measured by the post-operative CT scan.

SECONDARY OUTCOMES:
UPDRS (Unified Parkinson's Disease Rating Scale) Part III motor score | Week 15 to Week 40
  Changes in severity of PD (Parkinson's disease) motor symptoms assessed by UPDRS Part III motor scores
TUG (Timed Up and Go) test | Week 15 to Week 40
  Changes in mobility assessed by TUG test
UPDRS Total score (Part I-IV) | Week 15 to Week 40
  Change in severity of PD non-motor and motor symptoms assessed by UPDRS Part I-IV total scores (Parts I, II and IV in ON-state; Part III in OFF-state).
Home diary score | Week 16 to Week 24
  Change in functional status assessed by home diary score
PDQ-39 (Parkinson's Disease Questionnaire) score | Week 15 to Week 40
  Changes in health and daily activity assessed by PDQ-39 questionnaire score
change in CGI (Clinical Global Impressions) scale | Week 16 to Week 40
  • Change from baseline until end of treatment evaluation in mental status as measured by CGI scale.
Occurrence of blockage | Week 11 to Week 36
  Occurrence of blockage of implanted catheter preventing or limiting infusion assessed by measuring catheter pressure
Cessation of infusions | Week 11 to Week 36
  Cessation of infusions in an individual patient

OTHER OUTCOMES:
DAT (dopamine transporter)-PET imaging | Week 14 to Week 38
  Change in caudate and putamen DAT availability using PET imaging.
alpha-synuclein levels | Week 15 to Week 40
  Changes in serum and CSF (cerebrospinal fluid) concentrations of various α-synuclein species
Distribution of CDNF | Week 24 and Week 36
  Level of distribution of CDNF in serum and Cmax of CDNF in CSF
Daily activity measurement | Week 16 to Week 40
  Change in daily activity measured by Parkinson's KinetiGraph™ (PKG™) Data Logger
Coverage of infusate | Week 11 to Week 36
  Coverage of the infusate in target anatomy assessed by MRI (Magnetic resonance imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Per Svenningsson, MD, Principal Investigator — Karolinska University Hospital
Locations (3):
- Helsinki University Hospital, Helsinki, Finland
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Huddinge, Stockholm

IPD SHARING:
Plan to Share IPD: No